CLINICAL TRIAL: NCT02682836
Title: Physical Activity to Maintain Quality of Life and Physical Function in Women With Metastatic Breast Cancer: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC1537
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Breast Cancer
Keywords: physical activity; chemotherapy; fatigue
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Fatigue | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): Walk with Ease physical activity intervention
  Interventions: Behavioral: Walk with Ease

INTERVENTIONS:
Behavioral: Walk with Ease

SUMMARY:
Metastatic breast cancer (MBC) is an incurable disease. Maintaining optimum quality of life is a major goal of care. There is a strong body of evidence that exercise can reduce or manage fatigue, depression and insomnia in breast cancer patients; however, the evidence base is overwhelmingly in early stage cancer patients. The purpose of this study is to see if a home-based, self-directed walking program can have similar benefits in women with an MBC diagnosis. The primary objective is to evaluate whether engagement in physical activity will reduce fatigue during active treatment for MBC (baseline to 3 months); this is the primary endpoint. Secondary objectives pertain to feasibility of recruitment and retention of study participants and measuring changes between baseline, 3 months and 6 months in additional quality of life measures. Exploratory analyses pertain to changes in p16INK4a levels and sarcopenia between baseline and 3 months. The design is a single arm intervention trial in 30 patients. Findings from this study will provide preliminary data for a grant application to test the physical activity intervention in a randomized controlled trial (RCT) in a large sample of women with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 21 or older
* Metastatic breast cancer (MBC) diagnosis - Stage IV
* Receiving treatment regimen for MBC, but no more than 3 previous chemotherapy or biologic regimens
* Approval from the treating clinician to engage in moderate-intensity physical activity.
* Patient-assessed ability to walk and engage in moderate physical activity
* Proficient in English.
* IRB approved signed written informed consent.
* Willing and able to do all study requirements.

Exclusion Criteria:

* One or more significant medical conditions or other issues that in the physician's judgment preclude participation in the walking intervention.
* No more than 3 prior chemotherapy regimens.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
changes in fatigue scores | at 3 months
  Evaluate change in PROMIS Fatigue scores from baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten A Nyrop, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shachar SS, Heiling H, Muss HB, Meghan D, Wagoner CW, Deal AM, Nyrop KA. Physical Activity Intervention in Patients with Metastatic Breast Cancer During Active Treatment: Quality of Life and Function. Oncologist. 2023 Jan 18;28(1):84-e70. doi: 10.1093/oncolo/oyac232. PMID 36398879